CLINICAL TRIAL: NCT06402656
Title: Comparison of Customized and Standard Facemasks for Early Treatment of Class III Malocclusion: Randomized Crossover Study
Brief Title: Comparison of Customized and Standard Facemasks for Early Treatment of Class III Malocclusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LF14
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Malocclusion, Angle Class III; Extraoral Traction Appliances
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized facemask (Experimental)
  Interventions: Device: Customized facemask
- Standard facemask (Active Comparator)
  Interventions: Device: Standard facemask

INTERVENTIONS:
Device: Customized facemask — The customized face mask will be fabricated from a 3D digital image of the patient's face obtained by means of a 3D scanner. Such a scanner consists of 6 digital SLR cameras and software capable of processing a 3-D image of the patient's face exportable as an stl file.
  Arms: Customized facemask
Device: Standard facemask — The standard facemask is the commercially available Petit standard facemask
  Arms: Standard facemask

SUMMARY:
The aim of the study is to compare a customized facemask for the treatment of Class III malocclusion in the prepubertal growing patient (patients between the ages of 5 and 12 years) versus a standard commercial facemask. Specifically, preference, pain, difficulty in sleeping, time of use, and possible complications for the two types of facemasks will be analyzed.

This is a single-center, national, controlled, superiority, randomized, crossover, open-label study.

Each patient will be treated with both the customized facemask and the standard commercial facemask. Each patient will wear one type of facemask for 2 months and the other type of facemask for the next 2 months. After 2 weeks and at the end of therapy with each of the facemask types, the patient, with the possible help of the parents, will have to answer a questionnaire about pain and difficulty sleeping and report any complications. In addition, after completing both phases (fourth month), the patient should indicate a preference for one of the two types of mask with which to complete therapy for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 12 years;
* Class III malocclusion, for which early orthopedic treatment with rapid maxillary expander and facemask is indicated.
* signing of informed consent

Exclusion Criteria:

* Cleft lip and/or palate.
* Craniofacial syndromes.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire on the preference of the patient for one of the two types of face masks | 4 months
  The primary endpoint is a questionnaire on the preference between the two types of face masks at the end of the second phase of therapy (4 months after delivery of the first face mask)

SECONDARY OUTCOMES:
Pain reported by patients | At 2 weeks and at 2 months after delivery of each of the 2 face masks
  Pain measured through Visual Analogue Scale with minimum value of 0 and maximum value of 10. Higher scores mean worse pain.
Difficulty in sleeping reported by patients | At 2 weeks and at 2 months after delivery of each of the 2 face masks
  Difficulty in sleeping measured through VAS Visual Analogue Scale with minimum value of 0 and maximum value of 10. Higher scores mean more difficulty in sleeping.
Number of complications | At 2 weeks and at 2 months after delivery of each of the 2 face masks
  Number of complications
Total time wear | At 2 months after delivery of each of the 2 face masks
  Total time wear measured with a thermosensor (Theramon)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on appropriate request